CLINICAL TRIAL: NCT01444703
Title: Randomized, Double-blind Comparison of Licorice Versus Sugar-water Gargle for Prevention of Postoperative Sore Throat and Postextubation Coughing
Brief Title: Comparison of Licorice Versus Sugar-water Gargle for Prevention of Postoperative Sore Throat and Postextubation Coughing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, d sessler, Chairman, Outcomes Research Consortium, Outcomes Research Consortium
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 332/2010
Record Dates: First submitted 2011-09-23; First posted 2011-10-03 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Sore Throat
Keywords: Thoracic surgery; double-lumen endotracheal tube; intubation; extubation; sore throat; prevention of post-extubation sore throat
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sugar solution (Placebo Comparator): Gargle 5 minutes before induction of general anesthesia with sugar solution.
  Interventions: Other: sugar solution
- licorice (Active Comparator): Gargle 5 minutes before induction of general anesthesia with licorice solution.
  Interventions: Other: licorice solution

INTERVENTIONS:
Other: licorice solution — licorice (0.5 g)
  Arms: licorice
Other: sugar solution — sugar (5 g).
  Arms: sugar solution

SUMMARY:
The investigators propose to test the hypothesis that pre-operative gargling with licorice reduces the incidence of sore throat in rest after intubation with double-lumen endotracheal tubes compared to placebo after surgery through the first four post-extubation hours.

DETAILED DESCRIPTION:
Patients will be premedicated with up to 7.5 mg p.o. midazolam, per routine. They will be told that the study involves two different solutions for prevention of post-extubation sore throat.

Patients will be randomly assigned to gargle 5 minutes before induction of general anesthesia with: 1) licorice (0.5 g); or, 2) sugar (5 g). Randomization will be based on a computer-generated table of random numbers. Licorice or sugar (placebo) will be diluted in 30 ml water and filled in a small bottle by an independent apothecary of our university. All bottles will look similar and will not be opened until just before use. Investigator and patient will be blinded to the preparation used for gargle. Patients will be asked to gargle for two minutes, but not to swallow the solution.

General anesthesia will be induced with fentanyl ≈3 µg/kg, propofol ≈1.5 mg/kg, and rocuronium ≈0.6 mg/kg. Complete muscle relaxation will be confirmed by absence of palpable twitches in response to supra-maximal train-of-four stimulation of the ulnar nerve at the wrist. The trachea will then be intubated as gentle as possible. Intubation will be attempted with a Macintosh laryngoscope, but the anesthesiologists may subsequently use any other intubation equipment as necessary. Initial tube size will be 37 cm left in women and 39 cm left for men; however, other sizes can be used if clinically necessary. Endotracheal tube cuffs will be inflated with air to 20-25 mmHg as necessary to maintain an adequate seal.

General anesthesia will be primarily be maintained with sevoflurane. Patients lungs will be ventilated with O2 in air, usually with an inspired oxygen fraction (FiO2) of ≈40%. However, additional oxygen will be provided as clinically necessary, especially during one-lung ventilation. End-tidal CO2 will be maintained between 32 and 35 mmHg as clinically practical. Deep of anesthesia will be monitored by using bispectral index BIS, kept between 40 and 50. Small amounts of opioid will be permitted during surgery and in preparation for extubation. At the end of surgery, an intercostal plexus block -using up to 20 ml Ropivacaine 0.1% - will be performed by the surgeons. 1000 mg paracetamol will be given intravenously ten minutes before end of surgery. Post operative pain will be treated with fractional piritramid (Dipidolor) 3 mg IV as required.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic surgery with anticipated use of a double-lumen endotracheal tube;
* Anticipated extubation in the operating room;
* ASA Physical Status 1-3;
* Age 18- 90

Exclusion Criteria:

* Tracheal pathology, including tracheostomy;
* Surgery within the previous four weeks;
* Upper-respiratory tract infection;
* BMI higher exceeding 40 kg/m2;
* Known or suspected allergy to licorice;
* Use of non-steroidal anti-inflammatory drug medication within 24 hours;
* Chronic opioid use;
* Preoperative pain ≥ 2 on an 11-point Likert scale (0 = no pain; 10 = worst pain);
* Known or suspected difficult airway.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
sore throat in rest after intubation | up to 4 hours post-extubation
  We propose to test the hypothesis that pre-operative gargling with licorice reduces the incidence of sore throat in rest after intubation with double-lumen endotracheal tubes compared to placebo after surgery through the first four post-extubation hours.

SECONDARY OUTCOMES:
post-extubation coughing | up to four hours post-extubation
  Pre-operative gargling with licorice reduces sore throat pain during the initial postoperative day. Pre-operative gargling with licorice reduces the incidence of post-extubation coughing.
amount of coughing | 24 hours post operative
  Pre-operative gargling with licorice reduces the amount of coughing during the remainder of the first postoperative day.
sore throat in rest | first 24 hours after surgrey
  Pre-operative gargling with licorice reduces the incidence of sore throat in rest and during swallowing within the first 24 hours
incidence of sore throat during swallowing | first 24 hours after surgery
  Pre-operative gargling with licorice reduces the incidence of sore throat in rest and during swallowing within the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, MD, Study Chair — Outcomes Research Consortium, Cleveland Clinic
Locations (1):
- Universitätsklinik für Anästhesie, Intensivmedizin und Schmerztherapie an der medizinischen Universität Wien, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruetzler K, Fleck M, Nabecker S, Pinter K, Landskron G, Lassnigg A, You J, Sessler DI. A randomized, double-blind comparison of licorice versus sugar-water gargle for prevention of postoperative sore throat and postextubation coughing. Anesth Analg. 2013 Sep;117(3):614-621. doi: 10.1213/ANE.0b013e318299a650. Epub 2013 Aug 6. PMID 23921656